CLINICAL TRIAL: NCT01625195
Title: Causal Relationships Between LC-omega-3-enriched Diet and Cognition
Acronym: MOP201109
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRSC-2012
Record Dates: First submitted 2012-06-14; First posted 2012-06-21 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acid supplement (Placebo Comparator): This study will use a randomized placebo-controlled double-blind design and the intervention period will be 6 months. Participants will be instructed to consume 4 x 1285 mg fish oil capsules/d, two capsules with eachthe breackfast and two capsules with dinner. The daily treatment will provide 1.4 g/d of DHA and 1.8 g/d of EPA (Ocean Nutrition Canada, Dartmouth, NS). All capsules will contain orange flavor to mask the fishy taste and odor of the LC-omega-3 oil and will be provided to the participants monthly.
  Interventions: Dietary Supplement: omega-3 fatty acid supplementation
- Placebo (Active Comparator): This study will use a randomized placebo-controlled double-blind design and the intervention period will be 6 months. Participants will be instructed to consume 4 x 1285 mg capsules/d, two capsules with each of the main daily meals. The placebo will be composed of 50:50% corn/soybean oil as used in other randomized placebo-controlled trials.
  Interventions: Dietary Supplement: corn/soybean oil placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid supplementation — This study will use a randomized placebo-controlled double-blind design and the intervention period will be 6 months. Participants will be instructed to consume 4 x 1285 mg fish oil capsules/d, two capsules with each of the main daily meals. The placebo will be composed of corn/soybean oil as used in other randomized placebo-controlled trials. The daily treatment will provide 1.2 g/d of DHA and 2.4 g/d of EPA (Ocean Nutrition Canada, Dartmouth, NS). All capsules will contain citrus flavor to mask the fishy taste and odor of the LC-omega-3 oil and will be provided to the participants monthly.
  Other Names: MEG-3; 40/20 (EPA/DHA)ethyl esters fish oil capsules
  Arms: Omega-3 fatty acid supplement
Dietary Supplement: corn/soybean oil placebo — This study will use a randomized placebo-controlled double-blind design and the intervention period will be 6 months. Participants will be instructed to consume 4x 1285 mg capsules/d, two capsulesat breackfast and two capsules at dinner. The placebo will be composed of corn/soybean oil as used in other randomized placebo-controlled trials.
  Other Names: Meg-3 40:20 EPA:DHA ethyl esters
  Arms: Placebo

SUMMARY:
Nutrition is key to healthy aging for a number of diseases but the investigators have reported imbalances in the distribution of long chain omega-3 fatty acids (LC-omega-3) in the elderly and in the carriers of apolipoprotein E epsilon 4 (APOE4) isoform. Carrying APOE4 isoform is currently recognized as being the most important genetic risk factor of cognitive decline. The investigators believe that dysregulation of LC-omega-3 metabolism is intimately link with higher risk of cognitive decline. The current project will investigate whether there is a causal relationship between LC-omega-3-enriched diet and cognition using, on the one hand, a randomized double-blind placebo-controlled design and on the other hand, transgenic mice carrying human APOE4. In both study, the investigators will focus specifically on the distribution (level) of LC-omega-3 into lipoproteins with age and/or APOE4 isoform to evaluate whether dysfunctional transport of LC-omega-3 is associated with lower cognitive scores on visuospatial capacity, verbal fluency or working memory. In APOE4 mice, the investigators will evaluate LC-omega-3 brain uptake together with the level of LC-omega-3 in the brain membranes and the level of APOE protein within the brain. The present investigation will provide key basis for understanding how to develop nutritional strategies for healthy aging and the preservation of cognitive function.

DETAILED DESCRIPTION:
OVERALL AIM: In human and animal models, to investigate imbalances in the distribution of long chain omega-3 fatty acids (LC-omega-3) in plasma lipids and lipoproteins brought about by age and APOE4 genotype and to evaluate whether these imbalances are linked with cognitive functions. BACKGROUND: Risk of cognitive decline increases with age. Epidemiological studies strongly support a link between lower risk of cognitive decline and higher intake of fatty fish containing LC-omega-3. However, our clinical studies show that there are imbalances in the distribution of LC-omega-3 in plasma lipids that occur during aging and in the carriers of apolipoprotein E epsilon4 (APOE4) genotype, the most important genetic risk for cognitive decline. As a consequence, these imbalances appear to contribute to dysregulation of LC-omega-3 metabolism and to higher risk of cognitive decline. Our preliminary results in elderly humans show that visuospatial, verbal fluency and working memory scores are improved after 4 months supplementation with 3 g/d LC-omega-3, supporting a beneficial role of LC-omega-3 in cognition in the elderly. How this beneficial effect occurs is unknown but is potentially because the supplementation reverses or overrides imbalances in brain LC-omega-3 uptake and tissue content occurring during aging and in APOE4 carriers. Molecular mechanisms will be evaluated in 4-month and 15-month old transgenic mice expressing human APOE4. OVERALL HYPOTHESIS: Higher LC-omega-3 levels in lipoproteins are associated with higher LC-omega-3 brain uptake and membrane levels in APOE4 carriers leading to better cognitive scores on visuospatial, verbal fluency and working memory tests.

RESEARCH PLAN: Specific questions to be addressed are:

1) What is the role of APOE4 and blood lipoproteins on the causal relationship between a LC-omega-3-enriched diet and cognition? Three hundred participants aged between 20-80 y old will be recruited and randomized into a placebo (corn oil) or 3 g/d omega-3 fatty acid supplement for 6 months (150 subjects/group). LC-omega-3 use mostly VLDL and LDL to travel in the blood. Hence, we will collect blood samples once monthly for quantification of LC-omega-3 levels into VLDL, LDL and HDL, with longitudinal follow-up of LC-omega-3 throughout the supplementation period. This will provide key information regarding differences lipoprotein content of LC-omega-3 over the supplementation. We will perform cognitive tests with a focus on visuospatial, verbal fluency and working memory in the placebo and in the LC-omega-3 treated groups before and after the supplement. Age, sex and APOE4 genotype will be the interaction variables of interest. Statistical association test between cognitive scores and LC-omega-3 distribution in lipoproteins will also be performed to find the best LC-omega-3 marker associated with cognition.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged between 20-80 years old

Exclusion Criteria:

* tobacco use,
* malnutrition (assessed from blood albumin, hemoglobin and lipids),
* subjects taking an EPA+DHA supplement for more than one month,
* swallowing problems,
* severe gastro-intestinal problems,
* diabetes,
* uncontrolled thyroid disease,
* severe renal failure,
* liver disease or any other endocrine disorder,
* medication that would affect lipoprotein metabolism,
* chronic immune condition or inflammation (CRP > 10 mg/l, white cell count),
* cancer,
* recent major surgery or cardiac event,
* pregnant or lactating women,
* uncorrected visual or hearing problems,
* dementia,
* ongoing or past severe drug or alcohol abuse,
* psychiatric difficulties or depression, and
* ongoing or past intensive physical training

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in cognition | baseline and 6 months
  Evaluate change in visuospatial, verbal fluency or working memory with dietary intake (placebo or fish oil treatment.

SECONDARY OUTCOMES:
DHA level in plasma at baseline | baseline
  Evaluate DHA level in plasma lipids at baseline by age and by APOE genotype
Monthly DHA metabolism | once per month for 6 month
  Evaluate each month EPA and DHA level in plasma lipids and in lipoproteins

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Plourde, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- PL Léveillé, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
A description of the type of data required by other researchers will need approuval by Melanie Plourde. If biological samples are required by other researchers, they will need to get an ethical approuval by our research ethic committee.

REFERENCES:
- [Derived] Loukil I, Aguilera EC, Vachon A, Leveille P, Plourde M. Sex, Body Mass Index, and APOE4 Increase Plasma Phospholipid-Eicosapentaenoic Acid Response During an omega-3 Fatty Acid Supplementation: A Secondary Analysis. J Nutr. 2024 May;154(5):1561-1570. doi: 10.1016/j.tjnut.2024.03.013. Epub 2024 Mar 19. PMID 38513888